CLINICAL TRIAL: NCT03151122
Title: The Effect of Nurse-led Continuous Support Program on Neurodevelopment of Preterm Infants and Psychological Well-being of the Parents: A Randomized Controlled Trial
Brief Title: The Effect of a Nurse-led Continuous Support Program on Neurodevelopment of Preterm Infants
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Wuhan University (Other)
Responsible Party: Principal Investigator, Jun Zhang, Associate Professor, Wuhan University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2017-04
Record Dates: First submitted 2017-05-05; First posted 2017-05-12 (Actual); Last update posted 2020-05-20 (Actual); Status verified 2020-05

CONDITIONS: Preterm Infant
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- continuous care group (Experimental): continuous care group (CCG): This is the experimental group where continuous care supported would be offered by the nurse coordinated integrative health care team. which is, parents in this group receive support during infant hospitalization. The support covers both hospitalization phase and after-discharge phase. In-hospital support include educational support and promoting mother-infant attachment. Nurses will be responsible for home visits after infant discharge.
  Interventions: Behavioral: Nurse-led Continuous Support
- routine care group (Active Comparator): Routine Care Group (RCG): This is the comparison group of preterm infants. the routine care interventions generally include telephone reminding about follow-up care of the infants and hotline for parents to call when needed.
  Interventions: Procedure: routine follow-up care

INTERVENTIONS:
Behavioral: Nurse-led Continuous Support — The Nurse-Led Continuous Support was provided by a integrative care team. In-hospital support included(1) Promoting early parental-infant interaction;(2) Instruct the mother and/or father to use sensory stimulation activities to promote infant neuro-development in the NICU;(3) Parental educational support. The integrative care team will teach infant care skills, prepare them for successful transition from hospital to home setting.
  After infant discharge support will consist of regular home visits by the nurses. Home visits will be offered every other week until children reaching 3 Months of corrected age.
  Arms: continuous care group
Procedure: routine follow-up care — after infant discharge, parents were usually called upon to remind the date and time of follow-up care with physicians in outpatient department. A contact number was also given to parents in case they have questions about follow-up care.
  Arms: routine care group

SUMMARY:
The objective of the study is to establish a continuous nurse-led integrated support program and to exam its impact on preterm infant neurodevelopment.

Research hypotheses include:1. The continuous nurse-led integrated support will have significant impact on preterm infant neurodevelopment; 2.The support program will also have positive effect on parent psychological well-being.

DETAILED DESCRIPTION:
The objective of the study is to establish the continuous nurse-led integrated support program as well as exam its impact on neurodevelopmental health of preterm infants.

Research hypotheses:

1. Compared to control group, the preterm infants in the interventional group will experience significantly better performance on neuromotor, cognitive and social-emotional function at corrected age of 3 month;
2. In comparison with those receiving routine support, parents receiving nurse-led continuous support will have significantly higher parental self-efficacy and exhibited better psychological well-being;
3. Maternal parenting self-efficacy will mediate the relationship between nurse-led support and preterm infant neurodevelopment.

ELIGIBILITY:
Inclusion Criteria:

* Preterm infants born between 28-36 weeks of gestation;
* Parents residing in the same region for at least 5 years; .Parents agree to participate in the study.

Exclusion Criteria:

* infants with severe perinatal brain injury;
* infant with congenital anomalies

Ages: 28 Weeks to 36 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 140 (Estimated)
Dates: Start 2020-08-01 (Estimated); Primary Completion 2020-12-01 (Estimated); Study Completion 2021-04-01 (Estimated)

PRIMARY OUTCOMES:
Infant neuro-development assessed by the Ages and Stages Questionnaire (ASQ) | infant neuro-development will be measured at 3 months of corrected age.
  preterm infant will be assessed by the Ages and Stages Questionnaire (ASQ). The scale is used to help parent evaluate the development outcome of infants and young children by themselves.

SECONDARY OUTCOMES:
Maternal psychological well-being | assess when infants reach 1 month of corrected age.
  Edinburgh postnatal depression scale (EPDS) will be used to assess psychological well-being of preterm mothers.
Parental self-efficacy assessed by the Parenting Ladder Scale | assess when infants reach 3 month of corrected age
  The Parenting Ladder Scale will be used to determine the mothers/fathers' parental self-efficacy.

CONTACTS AND LOCATIONS:
Overall Officials: Chuan-Hua Yu, Study Chair — Wuhan University School of Health

IPD SHARING:
Plan to Share IPD: No